CLINICAL TRIAL: NCT05383339
Title: Biomarkers in Autoimmune Diseases, Vasculitis and Auto Inflammatory Diseases
Acronym: BIOMAI
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: APHP220486
Record Dates: First submitted 2022-05-09; First posted 2022-05-20 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Autoimmune Diseases; Vasculitis; Autoinflammatory Disease
Keywords: Autoimmune Diseases; Vasculitis; Autoinflammatory Disease; disease activity biomarkers cytokine and lymphocyte profile
MeSH Terms: conditions — Autoimmune Diseases; Vasculitis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Patients with autoimmune diseases, vasculitis and autoinflammatory diseases
  Interventions: Other: Blood collection

INTERVENTIONS:
Other: Blood collection — - 56mL blood collected additionally to routine care

SUMMARY:
The objective of this work is to identify, in patients with autoimmune diseases, systemic vasculitis and autoinflammatory disease, cytokine and lymphocyte biomarkers of activity of these diseases to identify follow-up biomarkers, in order to personalize the follow-up and the treatments for each patient.

Immunological data will be obtained from biological samples collected as part of the usual patient care pathway (Blood and tissues sampling) The study will take place in the Department of Internal Medicine and Clinical Immunology (DMIIC), that is certified as the National Reference Centre for Rare Systemic Autoimmune Diseases and the National Reference Centre for Inflammatory Autoinflammatory Diseases and Inflammatory Amyloidosis (CEREMAIA). Its objective is to contribute to the advancement of fundamental knowledge in immunology, in particular to develop prognostic biomarkers of the activity of autoimmune diseases, systemic vasculitis and autoinflammatory diseases by using blood tests.

DETAILED DESCRIPTION:
Autoimmune systemic diseases, systemic vasculitis and autoinflammatory diseases are diseases involving the innate and adaptive immune systems. The pro and anti-inflammatory cytokines, and the T and B lymphocytes appear as key actors of these pathologies, at the interface between the innate and adaptive immune system. The evolutionary profile of patients is highly variable, with some patients with minor forms mainly affecting the skin and joints for example, and others with potentially serious organ damage (e.g., renal involvement in lupus or vasculitis). At this time, we do not have markers to identify patients who will exhibit severe forms. Besides, treatments have evolved a lot over the years and mainly aime at controlling inflammation, either through non-target treatments (conventional immunosuppressants) or targeted biotherapies (anti-TNF, anti-interleukin 6, etc.). However, these treatments have in common to be suspensive in the majority of cases and the systemic diseases described tend to relapse frequently without clearly identifying clinical or biological factors predicting relapse. Patients are therefore exposed to treatments with many short-, medium- and long-term side effects without being able to identify precisely which patients benefit and which patients do not need further treatment.

The objective of this work is to identify, in patients with autoimmune diseases, systemic vasculitis and autoinflammatory disease, cytokine and lymphocyte biomarkers of activity of these diseases to identify follow-up biomarkers, in order to personalize the follow-up and the treatments for each patient.

Immunological data will be obtained from biological samples collected as part of the usual patient care pathway (Blood samples and tissues sampling) The Department of Internal Medicine and Clinical Immunology (DMIIC) is certified as the National Reference Centre for Rare Systemic Autoimmune Diseases and the National Reference Centre for Inflammatory Autoinflammatory Diseases and Inflammatory Amyloidosis (CEREMAIA). It has a fundamental research laboratory dedicated to the immunology of translational systems. Its objective is to contribute to the advancement of fundamental knowledge in immunology and in particular to develop prognostic biomarkers of the activity of autoimmune diseases, systemic vasculitis and autoinflammatory diseases by using blood tests. Several thousand patients with various autoimmune and autoinflammatory diseases are followed in the DMIIC, making the Department particularly suitable for this type of research.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 18 years of age or older
* Patients with autoimmune systemic disease, systemic vasculitis or autoinflammatory disease, defined by the international criteria in force for each pathology, among the following:

  * Connectivities: lupus, Sjögren syndrome, antiphospholipid syndrome, mixed connectivity and Sharp syndrome, scleroderma, myositis
  * Vasculitis of large, small and medium vessels: giant cell arteritis, Takayasu arteritis, Behçet disease, ANCA vasculitis, cryoglobulinemic vasculitis, IgA vasculitis (rheumatoid purpura)
  * Buerger's disease (obliterating thromboangitis)
  * Granulomatosis and sarcoidosis
  * Uveitis
  * Monogenic and polygenic autoinflammatory diseases: family Mediterranean fever, TRAPS, CAPS, chronic atrophic polychondritis, pericarditis
  * Recurrent fevers and unexplained inflammatory syndromes
  * Inflammatory amyloidosis
* Patients affiliated to French social security

Exclusion Criteria:

* Vulnerable populations:

  * Persons deprived of liberty by judicial or administrative decision;
  * Persons receiving psychiatric care without their consent;
  * Adult subject to a legal protection measure (guardianship, curatorship);
  * Persons unable to give their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with autoimmune diseases, systemic vasculitis and/or autoinflammatory disease
Sampling Method: Non-Probability Sample
Enrollment: 2250 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2031-11-29 (Estimated); Study Completion 2031-11-29 (Estimated)

PRIMARY OUTCOMES:
Correlation between cytokine and lymphocyte profile and disease activity | through study completion, an average of 9 years
  Identification of new biomarkers of the activity of autoimmune diseases, systemic vasculitis and autoinflammatory diseases, using flux cytometry and ELISA analysis.

SECONDARY OUTCOMES:
Characterization of new cytokines involved in these pathologies | through study completion, an average of 9 years
  Characterization of new cytokines involved in autoimmune diseases, systemic vasculitis and autoinflammatory diseases using ELISA analysis..
Characterization of new lymphocytes types involved in these pathologies | through study completion, an average of 9 years
  Characterization of new lymphocytes types involved in autoimmune diseases, systemic vasculitis and autoinflammatory diseases using flux cytometry analysis.
Correlation between the cytokine and lymphocyte profile, and the evolution of these pathologies (evolution towards mild forms, towards serious forms, death, frequency of relapses, etc.) | through study completion, an average of 9 years
  Determine predictive biomarkers of disease prognosis
Correlation between the cytokine and lymphocyte profile, and the clinical presentation of each pathology | through study completion, an average of 9 years
  Establish associations between different molecular subtypes, clinicohistological factors and main clinical signs.
Description of the cytokine and lymphocyte profile of each pathology. | through study completion, an average of 9 years
  Establish a molecular classification specific to each type of pathology: autoimmune diseases, systemic vasculitis and autoinflammatory diseases

CONTACTS AND LOCATIONS:
Overall Officials: David Saadoun, Professor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Département de Médecine Interne et Immunologie Clinique (DMIIC), Hôpital Pitié-Salpêtrière, Paris, France, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: website for Immunology Department of la Pitié Salpétrière hospital (Département de Médecine Interne et Immunologie Clinique) — http://www.maladiesautoimmunes.com/